CLINICAL TRIAL: NCT03435887
Title: Piloting At-birth Point of Care HIV Testing Strategies in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sarah Kessler, PhD, MPH, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00140399; R01HD076673-04S2 (NIH)
Record Dates: First submitted 2018-01-08; First posted 2018-02-19 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: Point of Care Testing; HIV; Pediatric HIV-exposed infants; at-birth testing; early infant diagnosis; Kenya
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alere q HIV-1/2 Detect for point of care infant testing (Active Comparator): POC testing with Alere q HIV-1/2 Detect at birth and 6-weeks postnatal in parallel with standard of care HIV DNA PCR testing
  Interventions: Behavioral: Alere q HIV-1/2 Detect for point of care infant testing; Behavioral: HIV DNA PCR testing (Standard of Care)
- GeneXpert HIV-1 Qual for point of care infant testing (Active Comparator): POC testing with GeneXpert HIV-1 Qual at-birth and at 6-weeks postnatal in parallel with standard of care HIV DNA PCR testing
  Interventions: Behavioral: GeneXpert HIV-1 Qual for point of care infant testing; Behavioral: HIV DNA PCR testing (Standard of Care)

INTERVENTIONS:
Behavioral: Alere q HIV-1/2 Detect for point of care infant testing — The investigators will pilot the Alere q HIV-1/2 Detect mobile system for point of care (POC) infant testing at two of the study hospitals. A blood sample will be collected from each HIV-exposed infants at birth (before discharge from Maternity or at first follow-up MCH visit within 14 days postnatal) and at 6-week EID visit (4-8 weeks postnatal) for analysis with Alere q HIV-1/2 Detect, with results available within 1-2 hours to enable mother notification at the same clinic visit.
  Arms: Alere q HIV-1/2 Detect for point of care infant testing
Behavioral: GeneXpert HIV-1 Qual for point of care infant testing — The investigators will pilot the GeneXpert HIV-1 Qual mobile system for point of care (POC) infant testing at two of the study hospitals. A blood sample will be collected from each HIV-exposed infants at birth (before discharge from Maternity or at first follow-up MCH visit within 14 days postnatal) and at 6-week EID visit (4 to <24 weeks postnatal) for analysis with GeneXpert HIV-1 Qual, with results available within 1-2 hours to enable mother notification at the same clinic visit.
  Arms: GeneXpert HIV-1 Qual for point of care infant testing
Behavioral: HIV DNA PCR testing (Standard of Care) — This is the standard of care for infant HIV testing. A dried blood spot sample will be collected from the infant and shipped to a central laboratory for HIV DNA PCR testing. Results will then be returned to the hospital.

SUMMARY:
Innovative strategies to expedite HIV diagnosis among exposed infants, including at-birth testing and two portable point-of-care (POC) diagnostic systems, will be piloted using an implementation framework. The programmatic impact of these tools on early infant diagnosis (EID) will be measured in comparison with parallel standard of care (SOC) HIV DNA PCR testing initiated at 6 weeks of age.

DETAILED DESCRIPTION:
Testing HIV-exposed infants by polymerase chain reaction (PCR) testing at 6 weeks is often not early enough to mitigate the substantial mortality peak that occurs around 2-3 months of age. Initial testing at birth would foster more rapid identification of infants with intrauterine (IU) infection and speed up the initiation of antiretroviral therapy (ART) for HIV-positive infants. Consequently, Kenya introduced new early infant diagnosis guidelines recommending at-birth (0-2 weeks) virologic testing in addition to the SOC tests at 6 weeks (6 - <24 weeks), 6 months and 12 months. POC testing performed in the clinic setting can potentially further reduce the time to diagnosis. Investigators will pilot test the implementation, performance, and cost-effectiveness of two POC test systems (Xpert HIV-1 Qual, Alere q HIV-1/2 Detect) in samples from neonates (at-birth test) and older infants (6-week test) in four government hospitals in Kenya.

In the formative phase of the study, interviews will be conducted with parents, providers and community members regarding benefits and concerns about the implementation of at-birth and POC testing. Interviews with parents (pregnant women living with HIV and their partners if available) will focus on the impact for the child and family. Interviews with providers who would carry out POC testing at each site (maternity nurses, mentor mothers, hospital laboratory staff) will highlight issues of training, logistics and implementation. Interviews with community members (parents of HIV-exposed infants, community health workers, community leaders) in surrounding communities will elicit attitudes and suggestions regarding the potential for POC HIV testing in hard to access communities. Investigators will develop a codebook with typical exemplars for each theme, calculating the frequency and distribution of themes within the larger topic areas. The study team will rapidly review themes to inform the POC pilot.

In the intervention phase the investigators will pilot at-birth and POC infant testing strategies in four hospitals over a continuous 12-month enrollment period. Sites will be randomized to pilot Xpert HIV-1 Qual (n=2) or Alere q HIV-1/2 Detect (n=2), both targeting the at-birth and 6-week testing points. A second blood sample will be collected at each time point to be tested by SOC laboratory-based HIV DNA PCR, which will correspond with the Kenya government's 2016 guidelines that recommend adding an at-birth test to the EID schedule. At-birth samples will ideally be collected within 24 hours of delivery and results communicated to the mother with counseling prior to discharge from maternity. The expected due dates of exposed infant will be tracked to encourage mothers who deliver outside the hospital to return for infant testing within two weeks postnatal. Infants enrolled in this pilot will be tracked until HIV results at birth and 6 weeks postnatal have been provided by POC and standard PCR, or until ART is initiated for HIV-positive infants. Investigators will assess user uptake, age at notification of HIV test results, age of ART initiation among HIV+ infants, POC machine performance, costs, and user experiences (providers will participate in a monthly focus group to discuss challenges and solutions) to inform the feasibility and optimal implementation of Kenya's 2016 at-birth test recommendation and of the mobile POC test systems for the improvement of EID outcomes.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive pregnant women enrolled in PMTCT services or who deliver at the study hospitals and/or mothers with exposed infants presenting for EID prior to 24 weeks
* Provide informed consent

Exclusion Criteria:

* HIV-positive pregnant women less than 18 years of age
* HIV-positive pregnant women unable to provide informed consent
* HIV-exposed infants presenting for HIV testing at > 24 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1999 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of infants tested at birth | 0-4 weeks
  The proportion of infants receiving HIV testing (POC and/or PCR) during the birth testing window
Proportion of infants tested at 6-weeks | 4-12 weeks postpartum
  The proportion of infants receiving HIV testing (POC and/or PCR) during the 6 week window

SECONDARY OUTCOMES:
Completeness of POC and SOC tests | up to 24 weeks postnatal
  Proportions of birth and 6-week tests with results returned and notified to mother
Efficiency of POC and SOC tests | up to 24 weeks postnatal
  Measures include turnaround time (TAT) associated with key steps in POC or SOC testing: TAT from specimen collection to result availability, TAT from result availability to mother notification of results, and overall TAT from specimen collection to mother notification.
Retention in EID services | up to 24 weeks postnatal
  Complete retention will be measured as the proportion of infants receiving a completed sequence of at-birth test result notification, 6-week-postnatal test result notification, and antiretroviral therapy (ART) initiation if HIV-positive.
POC system implementation | Month 12
  Number of POC tests performed successfully, versus indeterminate results or failed tests, on each platform.
  Number of missed opportunities to engage infants with POC testing due to documented machine breakdown, machine error, or cartridge stockout.
Costs | Month 12
  Costs of implementing each POC strategy into an existing system compared to HIV DNA PCR will be quantified, including up-front purchase of machines and accessory equipment; site-specific training and secure equipment storage; purchase of test cartridges, including delivery and customs fees; and machine repair.
Infant age at notification of HIV test results (birth and 6 week) | 0-8 weeks postnatal
  Infant age when mother is notified of at-birth (0-2 weeks postnatal) and 6 week (4-8 wks) POC and SOC test results

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kessler, PhD, Principal Investigator — University of Kansas Medical Center; Raphael Lwembe, PhD, Principal Investigator — Kenya Medical Research Institute
Locations (5):
- University of Kansas Medical Center, Kansas City, Kansas, United States
- Kenya (4):
  - Kisumu County Hospital, Kisumu
  - Kombewa District Hospital, Kombewa
  - Tudor Sub-County Hospital, Mombasa
  - Rift Valley Provincial General Hospital, Nakuru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandbulte MR, Gautney BJ, Maloba M, Wexler C, Brown M, Mabachi N, Goggin K, Lwembe R, Nazir N, Odeny TA, Finocchario-Kessler S. Infant HIV testing at birth using point-of-care and conventional HIV DNA PCR: an implementation feasibility pilot study in Kenya. Pilot Feasibility Stud. 2019 Jan 25;5:18. doi: 10.1186/s40814-019-0402-0. eCollection 2019. PMID 30701079
- [Result] Wexler C, Maloba M, Brown M, Mabachi N, Goggin K, Gautney B, Odeny B, Finocchario-Kessler S. Factors affecting acceptance of at-birth point of care HIV testing among providers and parents in Kenya: A qualitative study. PLoS One. 2019 Nov 22;14(11):e0225642. doi: 10.1371/journal.pone.0225642. eCollection 2019. PMID 31756242
- [Result] Wexler C, Kamau Y, Halder R, Brown M, Maloba M, Mabachi N, Sandbulte M, Gautney B, Goggin K, Odeny T, Finocchario-Kessler S. "Closing the Gap": Provider Recommendations for Implementing Birth Point of Care HIV Testing. AIDS Behav. 2019 Apr;23(4):1073-1083. doi: 10.1007/s10461-018-2363-3. PMID 30542834
- [Derived] Wexler C, Kamau Y, Muchoki E, Babu S, Maosa N, Maloba M, Brown M, Goggin K, Mabachi N, Gautney B, Finocchario-Kessler S. Implementing at-birth, point-of-care HIV testing in Kenya: a qualitative study using the Consolidated Framework for Implementation Research. Implement Sci Commun. 2021 Aug 11;2(1):89. doi: 10.1186/s43058-021-00188-9. PMID 34380567